CLINICAL TRIAL: NCT04327362
Title: TDCS-Augmented Prolonged Exposure Therapy for PTSD: a Multiple Baseline Within-Subject Clinical Trial
Brief Title: TDCS-Augmented Prolonged Exposure Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn due to delay in recruitment due to COVID-19; the PI also moved to a new institution.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00093774
Record Dates: First submitted 2020-03-25; First posted 2020-03-31 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Posttraumatic Stress Disorder; PTSD; Anxiety; Depression
Keywords: Non-invasive brain stimulation; Transcranial direct current stimulation; Exposure therapy; Prolonged Exposure; Civilians; Veterans; Trauma; Posttraumatic stress disorder; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; Wounds and Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned following stratification by baseline severity of PTSD symptoms, medication status, and sex to one of five clusters defined by the point of cross-over from sham to active tDCS administered just prior to PE therapy sessions, with the earliest cross-over occurring at session 4, and the latest at session 8.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Customized software involving use of a coding scheme will be used to allow complete blinding to whether active or sham tDCS is administered. The participants, tDCS administrators, therapists, and outcome assessors will remain blind to tDCS condition. The integrity of blinding procedures will be evaluated by self-report questionnaires administered at each treatment visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Cluster 1: Sham to active tDCS crossover at PE Session 4. (Experimental): Participants in this cluster will receive 20 min. of sham tDCS prior to the PE sessions 1-3, and 20 min. of active tDCS prior to PE sessions 4-10.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Prolonged Exposure Therapy
- Cluster 2: Sham to active tDCS crossover at PE Session 5. (Active Comparator): Participants in this cluster will receive 20 min. of sham tDCS prior to the PE sessions 1-4, and 20 min. of active tDCS prior to PE sessions 5-10.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Prolonged Exposure Therapy
- Cluster 3: Sham to active tDCS crossover at PE Session 6 (Active Comparator): Participants in this cluster will receive 20 min. of sham tDCS prior to the PE sessions 1-5, and 20 min. of active tDCS prior to PE sessions 6-10.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Prolonged Exposure Therapy
- Cluster 4: Sham to active tDCS crossover at PE Session 7. (Active Comparator): Participants in this cluster will receive 20 min. of sham tDCS prior to the PE sessions 1-6, and 20 min. of active tDCS prior to PE sessions 7-10.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Prolonged Exposure Therapy
- Cluster 5: Sham to active tDCS crossover at PE Session 8. (Active Comparator): Participants in this cluster will receive 20 min. of sham tDCS prior to the PE sessions 1-7, and 20 min. of active tDCS prior to PE sessions 8-10.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Participants will receive 20 min. of either sham or active tDCS prior to PE sessions using a 1 x 1 tDCS device with a ring electrode configuration that allows relatively excitatory and focal stimulation of the dorsomedial prefrontal cortex (dmPFC). Electrodes consist of sponges in a silicone rubber holder with a metal mesh conductor saturated with normal saline. A center anode (2.5 cm diameter) and a ring-shaped cathode (diameter inner/outer: 9.2/11.50 cm) will be centered over the dmPFC, with the anode placed the midline at 15% of the Fz to FPz distance. Active stimulation will commence with a 15 sec. ramping up period to target current (1.5 mA), followed by constant current for 20 min., and a 15 sec. ramping down period. For all sham sessions, stimulation will be immediately ramped down over a 15 sec. period following the initial ramping up period, and subsequently ramped up over 15 sec. prior to the final ramping down period.
  Other Names: Soterix Medical 1 x 1 Transcranial Electrical Stimulator (tES)
Behavioral: Prolonged Exposure Therapy — All participants will receive 10 weekly sessions of standard Prolonged Exposure Therapy, or PE, which is a gold standard trauma-focused cognitive behavioral treatment for PTSD. The first sessions (1-2) predominately consist of psychoeducation about PTSD and the rationale for treatment, whereas subsequent sessions (3-10) consist of imaginal and in vivo exposure, involving repeated, prolonged, systematic, and deliberate practice approaching trauma reminders, as well as cognitive and emotional processing reactions to an index trauma memory.
  Other Names: PE; CBT; Trauma-focused therapy

SUMMARY:
The purpose of this study is to determine the effects of a brain stimulation technique known as transcranial direct current stimulation, or tDCS, on the benefits of Prolonged Exposure therapy, or PE, which is an effective treatment for posttraumatic stress disorder, or PTSD. tDCS has been demonstrated to be safe and effective for influencing brain activity by passing a weak electrical current through the scalp. In this study, tDCS is provided in addition to PE treatment, through the National Crime Victim's Research and Treatment Center at MUSC, or the PTSD Clinical Team Clinic within the Ralph H. Johnson VA Medical Center.

DETAILED DESCRIPTION:
This project implements a multiple baseline within-subject clinical trial design aiming to test whether tDCS targeting excitation of the medial prefrontal cortex (mPFC) can enhance a standard course of PE in a sample of adult civilians and Veterans (ages 18-65) who meet full DSM-5 criteria for chronic PTSD (i.e., > 3 months post-trauma; N = 20). All participants will receive a total of ten 60-min. sessions of manualized PE, preceded by 20 min. of either active or sham HD-tDCS. The stepped-wedge multiple baseline design features tDCS as a 2-level within-subject factor (Sham tDCS+PE vs. Active tDCS+PE), and between-subject comparisons based on stratified random assignment to cross-over from sham to active tDCS just prior to sessions 4 through 8. Strata will be defined by dichotomous classifications of possible confounds, including baseline severity (moderate vs. severe), psychotropic medication status (no vs. yes), and sex (female vs. male). The sample will consist of treatment-seeking civilian and Veteran participants referred by either of two of our consortium sites, including the National Crime Victim's Research and Treatment Center (NCVC) at MUSC, or the PTSD Clinical Team (PCT) at the Ralph H. Johnson VAMC, as well as community participants who respond to study advertisements.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65.
* Fluent in English.
* Diagnosis of chronic PTSD based on MINI for DSM-5 (> 3 mo. post-trauma)
* For Veterans recruited at the Ralph H. Johnson VA only: eligible to receive PE in the PCT clinic.

Exclusion Criteria:

* Currently receiving psychotherapy for another anxiety- or stress-related condition.
* Unstable dose of psychotropic medications within 6 weeks prior to baseline assessment
* Medical condition that would contraindicate participation in treatment or assessment activities (e.g., severe cardiovascular problems).
* Pregnancy
* Current severe major depressive disorder
* Current, or history of bipolar disorder
* Current, or history of psychotic symptoms
* Serious suicidal risk
* Active neurological conditions, e.g., seizures, stroke, loss of consciousness or concussion
* Contraindications for tDCS:
* Metal in the head.
* Implanted brain medical devices.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Clinician-Rated PTSD Symptom Severity | Pre-treatment (baseline), post-treatment (12 weeks post-baseline), and 1-month follow-up (16 weeks post-baseline)
  Clinician-administered PTSD Symptom Scale Interview for DSM-5 (PSSI-5).
  Total scores range from 0 to 80, with higher scores indicating greater severity of PTSD symptoms.
Change in Self-Reported PTSD Symptom Severity | Pre-treatment (baseline), post-treatment (12 weeks post-baseline), and 1-month follow-up (16 weeks post-baseline)
  Self-report scores on the PTSD Symptom Checklist for DSM-5 (PCL-5)
  Total scores range from 0 to 80, with higher scores indicating greater severity of PTSD symptoms.
Change in Self-Reported Post-traumatic Cognitions | Pre-treatment (baseline), post-treatment (12 weeks post-baseline), and 1-month follow-up (16 weeks post-baseline)
  Self-report scores on the Post-traumatic Cognitions Inventory (PTCI-9)
  Total scores range from 9 to 63, with high scores indicating greater endorsement of common and problematic trauma-related beliefs.
Change in Depression Symptoms | Pre-treatment (baseline), post-treatment (12 weeks post-baseline), and 1-month follow-up (16 weeks post-baseline)
  Self-report scores on the Beck Depression Inventory, 2nd Edition (BDI-II)
  Total scores range from 0 to 63, with higher scores indicating greater severity of depression symptoms.
Change in Anxiety Symptoms | Pre-treatment (baseline), post-treatment (12 weeks post-baseline), and 1-month follow-up (16 weeks post-baseline)
  Self-report scores on the Beck Anxiety Inventory (BAI)
  Total scores range from 0 to 63, with higher scores indicating greater severity of anxiety symptoms.

SECONDARY OUTCOMES:
Within- and Between-Session Change in Trauma-Related Emotional Distress | During weekly therapy sessions 1-10, for 10 weeks from baseline.
  Self-reported in-session Subjective Units of Distress Scale (SUDS)
  Peak distress among repeated ratings obtained during therapy sessions from 0 = "no distress" to 100 = "extreme distress". Ratings will be obtained up to 13 times at each weekly Prolonged Exposure therapy session, for 10 weeks.
Within- and Between-Session Change in Heart Rate | During weekly therapy sessions 1-10, for 10 weeks from baseline.
  Continuously recorded in-session heart rate
  Heart rate will be continuously recorded during each weekly Prolonged Exposure therapy session, for 10 weeks.
Within- and Between-Session Change in Physiological Activation | During weekly therapy sessions 1-10, for 10 weeks from baseline.
  Continuously recorded in-session skin conductance levels
  Skin conductance levels will be continuously monitored during each weekly Prolonged Exposure therapy session, for 10 weeks.
Between-Session Change in Trauma Memory Engagement and Emotional Processing | During weekly therapy sessions 1-10, for 10 weeks from baseline.
  Therapist-report scores on the Prolonged Exposure Therapist Questionnaire
  Total scores range from 0 to 35, with higher scores indicating greater retrieval, processing, and meaning making during imaginal revisiting of the index trauma memory.

CONTACTS AND LOCATIONS:
Overall Officials: Adam R. Cobb, Ph.D., Principal Investigator — Medical University of South Carolina & Ralph H. Johnson VAMC Consortium; Lisa M. McTeague, Ph.D., Principal Investigator — Medical University of South Carolina & Ralph H. Johnson VAMC Consortium; Bethany C. Wangelin, Ph.D., Principal Investigator — Medical University of South Carolina & Ralph H. Johnson VAMC Consortium
Locations (1):
- National Crime Victim's Research & Treatment Center, Department of Psychiatry and Behavioral Sciences, Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No